CLINICAL TRIAL: NCT06171321
Title: Circulating Tumor DNA Guided Adjuvant Chemotherapy for Biliary Tract Carcinoma: A Prospective Clinical Trial
Brief Title: Circulating Tumor DNA Guided Adjuvant Chemotherapy for Biliary Tract Carcinoma
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai East Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: [2023] R&R No. (107)
Record Dates: First submitted 2023-11-14; First posted 2023-12-14 (Actual); Last update posted 2023-12-14 (Actual); Status verified 2023-11

CONDITIONS: Biliary Tract Cancer
Keywords: S-1; circulating tumor DNA (ctDNA)
MeSH Terms: conditions — Biliary Tract Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: Patients testing negative for ctDNA treated using standard of care treatment (No Intervention): Postoperative ctDNA-negative patients receive oral Teysuno (S-1) for adjuvant therapy。
- Group 2: Patients with a positive ctDNA test are treated with an escalation strategy (Experimental): Postoperative ctDNA-positive patients receive intravenous combined oral Teysuno (S-1) for adjuvant therapy。
  Interventions: Drug: S-1(Intravenous combined with oral)

INTERVENTIONS:
Drug: S-1(Intravenous combined with oral) — Oral combined with intravenous S-1 for ctDNA-positive patients (escalating treatment strategy)
  Arms: Group 2: Patients with a positive ctDNA test are treated with an escalation strategy

SUMMARY:
In recent years, circulating tumor DNA (ctDNA)had achieved encouraging results in monitoring recurrence and metastasis after surgery, and has potential clinical application value. The presence of ctDNA after surgery predicts very poor recurrence-free survival, whereas its absence predicts a low risk of recurrence. The benefit of adjuvant chemotherapy for ctDNA-positive patients is not well understood.

DETAILED DESCRIPTION:
The results of the PRODIGE-12/ACCORD-18 study showed that, with a median follow-up of 47 months, the adjuvant chemotherapy arm did not lead to a significant improvement in recurrence-free survival (RFS) and overall survival (OS). Notably, the patients with gallbladder cancer experienced adjuvant chemotherapy significantly worse RFS and OS compared to those in the monitoring arm. ctDNA risk stratifies patients to guide adjuvant treatment decisions This study aimed to demonstrate that a escalation strategy of ctDNA guided adjuvant chemotherapy is superior to standard of care treatment as measured by 2 year disease free survival (DFS) in patients with stage II- III biliary tract cancers with minimal residual disease (MRD) (ctDNA positive).

ELIGIBILITY:
Inclusion Criteria:

* 1) Patients with pathologically confirmed BTCs according to the UICC/AJCC TNM staging system (8th edition 2017) for stage II-III tumours. Patients eligible for radical resection of BTCs. No synchronous or metastatic malignant tumour found in other organs other than the primary tumor.

  2) Personal status (PS) score as over 80 or Eastern Cooperative Oncology Group (ECOG) score as 0 ~ 2.

  3）With expected survival of more than 12 months. 4) Radical operation performed.

Exclusion Criteria:

* 1) Patients with positive surgical margins and residual lesions after biliary tract tumor surgery.

  2) Blood transfusion performed during operation or within 2 weeks before operation.

  3) Have a history of other malignant tumors within 5 years.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2023-12 (Estimated); Primary Completion 2025-11-15 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
ctDNA guided adjuvant chemotherapy versus Translational sub study | Up to 60 months
  To demonstrate the superiority of an escalation strategy of ctDNA-guided adjuvant chemotherapy over standard-of-care treatment, 2-year disease-free survival (DFS) was measured as 2-year Disease-Free Survival (DFS) in high-risk stage II-III BTC patients with no evidence of minimal residual disease (ctDNA-negative).
Sensitivity of postoperative ctDNA in monitoring recurrence and metastasis | Up to 60 months
  Number of patients with ctDNA positive and imaging confirmed recurrence or metastasis / number of all imaging confirmed recurrence or metastasis
Specificity of postoperative ctDNA in monitoring recurrence and metastasis | Up to 60 months
  Number of patients with ctDNA negative and no recurrence and metastasis confirmed by imaging / number of patients with no recurrence and metastasis confirmed by imaging
Accuracy of postoperative ctDNA in monitoring recurrence and metastasis | Up to 60 months
  True positive/ctDNA-positive samples

SECONDARY OUTCOMES:
overall survival (OS) | From date of randomization until the date of first documented date of death from any cause, assessed up to 60 months.
  Overall survival of included patients
ctDNA clearance rate | Up to 60 months
  The rate of ctDNA positive before chemotherapy that turns negative after adjuvant chemotherapy

CONTACTS AND LOCATIONS:
Locations (1):
- East Hospital, Tongji University School of Medicine, Shanghai, China